CLINICAL TRIAL: NCT05926115
Title: Phenotype and Epidemiology of the Polycystic Ovary Syndrome (PCOS) in Colombia (PEP - Colombia) Study.
Acronym: PEP-Colombia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto de fertilidad humana, InSer (Other)
Collaborators: University of Alabama at Birmingham (Other); Colmédicos S.A.S. (Unknown); ABAD Laboratorio (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1006
Record Dates: First submitted 2023-06-01; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Polycystic Ovary Syndrome; Hyperandrogenism; Endocrine System Diseases
Keywords: Polycystic Ovary; Hyperandrogenism; Hirsutism; Oligomenorrhea; Anovulation; Menses, Irregular
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism; Endocrine System Diseases; Hirsutism; Oligomenorrhea; Anovulation; Menstruation Disturbances | interventions — Ultrasonography; Hematologic Tests

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Ultrasound — During the initial visit, a transvaginal or transabdominal pelvic ultrasonography will be performed in all participants, based on the sexual history and consent form by trained gynecologists who are part of study investigators. A transvaginal ultrasound is the accepted and validated method to assess the ovarian morphology in the study of patients with PCOS.
  Other Names: Pelvic ultrasound
Diagnostic Test: Venous puncture — After an overnight fast of at least 6 hours (ideally), a 18 ml sample of venous blood will be collected from each study participant (i.e., the basal fasting sample). About 12 ml of the venous blood will be collected in plain tubes for serum cryopreservation and subsequent analysis, and the remainder in plain tubes for immediate glucose estimation in serum.
  Other Names: Blood test

SUMMARY:
The goal of this observational study is to know the prevalence of PCOS among economically productive and reproductive age women from Medellín and the Valle de Aburrá, Colombia. The main questions it aims to answer are:

1. What is the phenotypic distribution of PCOS detected in women seeking medical attention as a requirement for employment in Medellín and the Valle de Aburrá, Colombia?
2. What is the effect of environmental factors, such as geographical location and diet, and biological factors (such as obesity and ethnicity/race) on the prevalence and phenotype of PCOS in this populatión?

Participants will undergo anthropometric measurements and physical examination for hirsutism, acne, alopecia, acanthosis nigricans, and thyroid enlargement. During the initial visit, a transvaginal or transabdominal pelvic ultrasonography will be performed. A sample of venous blood will be collected in plain tubes for serum cryopreservation and for immediate glucose estimation. Some participants will be rescheduled for a second evaluation visit for additional assessment when they have a possible PCOs.

DETAILED DESCRIPTION:
During the first visit, potential study participants, scheduled for routine occupational pre-admission medical examination at Colmédicos Medical Centre, will be invited to participate in the study. Eligible study participants will be counselled on the objectives of the study and the study protocol and a copy of the consent form will be handed to them. A confidential study register containing details of potential study participants (name, age, height, weight, and contact) will be start on the first visit day. Informed written consent will be obtained from each study participant before recruitment for the study in the evaluation visit number one. All study participants personal data will be protected according to the law (ley 1581de Colombia).

1. Evaluation Visit #1:

   After obtaining an informed consent, data will be collected from each study participant using a standard format in a clinical report form (CRF) for uniform data collection from all participants. Each CRF will bear a unique serial identification number and will be written in the local language. The CRF will be filled by a trained researcher (including the PI, co-investigators and medically trained research assistants). All CRF will be checked for missing data within 24 hours of completion, and any missing data will be detected and collected immediately. At no time, will the study personnel have access to the participant´s medical occupational records, following the restrictions defined in the colombian legislation (resolution 2346 de 2007, R 1918 de 2011).

   Each participant will undergo anthropometric measurements (weight, height, waist circumference and hip circumference) and physical examination for hirsutism, acne, alopecia, acanthosis nigricans, and thyroid enlargement. Participants with an initial hirsutism (mFG) score of 4 or more (≥ 4) will be re-assessed by a physician. During the initial visit at Colmédicos, a transvaginal or transabdominal pelvic ultrasonography will be performed in all participants, based on the sexual history and consent form by trained gynecologists who are part of study investigators. A transvaginal ultrasound is the accepted and validated method to assess the ovarian morphology in the study of patients with PCOS.

   After an overnight fast of at least 6 hours (ideally), a 18 ml sample of venous blood will be collected from each study participant (i.e., the basal fasting sample). About 12 ml of the venous blood will be collected in plain tubes for serum cryopreservation and subsequent analysis, and the remainder in plain tubes for immediate glucose estimation in serum.
2. Sample Processing:

   The initial blood specimens will be labeled with the participant´s unique ID number, time and date of blood collection and date of last menstrual period (LMP). The samples will be obtained by trained laboratory personnel from Colmédicos medical center during the morning hours (08:00 to 10:00 hours), regardless of the participant's menstrual cycle. Participants with oligomenorrhoea or amenorrhoea will have a urine pregnancy done test prior to blood sampling.

   At Colmédicos laboratory, the blood samples will be separated into serum, plasma and whole blood by centrifugation for 20 minutes at 3000 rpm. The biological specimens will be stored, in small aliquots (of 1,25 ml), in 1.5 to 2.0 ml plastic containers (about 4 cryovials) able to withstand temperatures of -80 degrees centigrade. The aliquoted samples will be sent to the ABAD Zona 2 SUR laboratory (Carrera 32 No. 2 Sur 47 local 9701) in dry ice containers by the laboratory's courier staff where they will be stored at -20 degrees centigrade for a maximum of 3 months for processing. If necessary, for longer storage, the samples will be transferred to the Inser Medellin laboratory and stored at -80 degrees centigrade where they will remain in custody until their use or final disposal according to the established institutional waste management protocol.
3. Hormonal & chemical analyses:

   Samples for hormonal assay and the initial evaluation will be batched at regular intervals for the analysis every week to provide the study participants with timely results, allow classification of participants and minimize the impact of inter-assay variability. In addition, this will allow us to timely contact participants who require additional studies.

   All participants will be evaluated in a uniform manner regardless of the phase of the cycle in which they are.
4. Evaluating subjects with "Possible PCOS":

   The cohort of participants who initially meet clinical features suggestive of PCOS (i.e., HA, OA or PCOM, will be designated as "Possible PCOS", and will undergo the following measurements in their samples:
   1. In all "Possible PCOS" subjects TSH, prolactin (PRL), and 17-HP will be measured in the basal serum samples as well as fasting glucose.

      Note: All subjects diagnosed with PCOS should have a normal TSH, PRL, and 17-HP (basally or after acute ACTH stimulation).
   2. In women presenting clinically with HA+OA, if the TV-U/S performed demonstrates PCOM the subject is classified as having PCOS phenotype A (HA+OA+PCOM); if not the subject is classified as having PCOS phenotype B (HA+OA).
   3. Subjects presenting clinically with HA only will return during the luteal phase (days 21-24) of their menstrual cycle for a serum progesterone (P4) level. Subjects with HA who demonstrate OA (i.e., luteal P4 < 3 ng/mL) will be classified as having PCOS phenotype A if they have PCOM by TV-U/S (HA+OA+PCOM) or PCOS phenotype B (HA+OA) if they do not exhibit PCOM. HA subjects who also demonstrate PCOM, but no OA (i.e., luteal P4 ≥3 ng/mL) will be classified as PCOS phenotype C. Participants with HA, but no PCOM or OA will be classified as having isolated HA.
   4. Subjects presenting clinically with OA only, their basal serum samples will be assayed for androgen levels (total [TT] and free testosterone [FT], dehydroepiandrosterone sulphate [DHEAS], and androstenedione [A4]). Subjects with OA who demonstrate HA (i.e., elevated androgen levels) will be classified as having PCOS phenotype A if they have PCOM by TV-U/S (HA+OA+PCOM) or PCOS phenotype B (HA+OA) if they do not exhibit PCOM. OA subjects who also demonstrate PCOM, but no HA (i.e., normal androgen levels) will be classified as PCOS phenotype D. Participants with OA, but no PCOM or HA will be classified as having isolated OA.
   5. Subjects presenting with PCOM by TV-U/S will return during the luteal phase (days 22-24) of their menstrual cycle for a serum progesterone (P4) level and their basal serum samples will be assayed for androgen levels (total [TT] and free testosterone [FT], dehydroepiandrosterone sulphate [DHEAS], and androstenedione [A4]). Subjects with PCOM who demonstrate OA (i.e., luteal P4 < 3 ng/mL) will be classified as having PCOS phenotype D. If they also demonstrate HA (i.e., elevated androgen levels) (HA+OA+PCOM) will be classified as having PCOS phenotype A. PCOM subjects who also demonstrate HA, but no OA (i.e., luteal P4 ≥3 ng/mL) will be classified as PCOS phenotype C. Participants with PCOM, but no HA or OA will be classified as having isolated PCOM.
5. Diagnosing PCOS:

   Related or mimicking disorders will be excluded using history, physical examination, and serum TSH, PRL and 17-OHP. Study participants with a basal 17-OHP >2 ng/ml (or 200 ng/dl) will undergo a repeat 17-OHP measurement in the follicular phase and if the 17-OHP is still > 2ng/mL an acute adrenocorticotrophic hormone (ACTH) stimulation test will be performed to exclude non-classical congenital adrenal hyperplasia (NCAH). We estimate, considering our previous data, that approximately 6% of subjects screened will require an acute ACTH stimulation test.

   Overall, PCOS will be diagnosed when subjects present with either HA+OA+PCOM (phenotype A), HA+OA (phenotype B), HA+PCOM (phenotype C) and OA+PCOM (phenotype D) and demonstrate normal levels of TSH (0,37 to 4,7 mUI/L), PRL (<25 ng/mL) and 17-OHP, per our diagnostic algorithm.
6. Evaluation visit #2:

   In the following cases subjects will be rescheduled for a second evaluation visit (evaluation visit #2) for additional assessment:
   1. All subjects with PCOS will be scheduled for a return visit to undergo a 2-hour 75g oral glucose tolerance test (OGTT) with 3 ml of venous blood collected in serum tubes at 0 minutes and at 120 minutes post-glucose load. Glucose and insulin (from serum tubes) levels will be assessed at 0 and 120 min.
   2. Participants will be reevaluated during the follicular phase of the menstrual cycle (between day 1 and 5):

   i. With a repeat ultrasound in case there is a dominant follicle (≥ 10 mm) or an ovarian cyst at the initial ultrasound evaluation.

   ii. A repeat 17-hydroxyprogesterone (17-OHP) measurement in the event the initial 17-OHP is >2 ng/mL and was obtained during the luteal phase according to menstrual history. Approximately 50% of Participants evaluated in luteal phase are expected to have a 17-OHP >2 ng/mL.

   iii. An acute intravenous (iv) ACTH-1-24 (0.25 mg) stimulation test, if the initial and repeat 17-OHP obtained during the follicular phase, according to menstrual history, is > 2 ng/mL.
7. Reassessing hormonal levels:

At the completion of the study, a repeat analysis of the samples for androgen levels in all PCOS subjects and a group of 'super-controls' (30 controls) will be performed at a reference laboratory. A fasting glucose level also be analyzed in a group of super controls (100 controls). Genetic analysis could be performed depending on the availability of financial support in a reference laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 45 years.
2. Participants with thyroid dysfunction on medication will be included only if their TSH level is normal (prior to or at re-evaluation)
3. Participants with hyperprolactinemia will be included only if their prolactin (PRL) level is normal (prior to or at re-evaluation) b) Exclusion criteria

a. Women who are pregnant at the time of evaluation b. Postmenopausal women

Exclusion Criteria:

1. Women who are pregnant at the time of evaluation
2. Postmenopausal women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — PCOS is a female disorder
Study Population: Women seeking medical attention at Colmédicos medical center as a requirement for employment in Medellín and the Valle de Aburrá, Colombia.
Sampling Method: Non-Probability Sample
Enrollment: 626 (Estimated)
Dates: Start 2023-03-04 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of PCOS | Six months
  Prevalence of PCOS among a medically unselected population-based sample representing the Latino population. In addition, Percentage of participants with phenotype A, B, C or D, among participants diagnosed with PCOS.

SECONDARY OUTCOMES:
Percentage of participants with obesity, endocrine disorders, metabolic syndrome, hyperandrogenism, hirsutism, oligomenorrhea, anovulation and irregular menses | Six months
  Percentage of participants with obesity, endocrine disorders, metabolic syndrome, hyperandrogenism, hirsutism, oligomenorrhea, anovulation and irregular menses among the study population, which will also have a detailed description of their demographic characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Azziz, M.D., Study Director — University of Alabama at Birminghan
Locations (1):
- Colmédicos S.A.S, Sabaneta, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No